CLINICAL TRIAL: NCT00906828
Title: Pharmacokinetics of Levodopa in Patients With Parkinson's Disease Treated With Levodopa/Carbidopa Infusion With and Without Oral COMT Inhibitors
Brief Title: Pharmacokinetics of Levodopa/Carbidopa Infusion With and Without Oral Catechol-O-methyl Transferase (COMT) Inhibitors
Acronym: DuoCOMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish Parkinson's Disease Foundation (Unknown); Swedish Society for Medical Research (Other)
Responsible Party: Dag Nyholm, MD, PhD, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DuoCOMT
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Parkinson Disease
Keywords: Levodopa/carbidopa infusion; entacapone; tolcapone; efficacy; pharmacokinetic; pharmacodynamics
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; entacapone; Tolcapone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. Duodopa, optimised dose (Active Comparator)
  Interventions: Drug: levodopa/carbidopa
- 2. 80% Duodopa + entacapone (Experimental): 80% of optimised Duodopa dose + two tablets of entacapone at t=0 hours and at t= 6 hours
  Interventions: Drug: entacapone
- 3. 80% Duodopa + tolcapone (Experimental): 80% of optimised Duodopa dose + two tablets of tolcapone at t=0 hours and at t= 6 hours
  Interventions: Drug: tolcapone

INTERVENTIONS:
Drug: levodopa/carbidopa — intestinal gel, continuous infusion (daytime or 24-hour)
  Other Names: Duodopa
  Arms: 1. Duodopa, optimised dose
Drug: entacapone — Tablet, 200 mg, given twice during the study at t=0h and t=5hrs
  Other Names: Comtess, Comtan.
  Arms: 2. 80% Duodopa + entacapone
Drug: tolcapone — Tablet, 100 mg, given twice during study, at t=0h and t=5hrs.
  Other Names: Tasmar
  Arms: 3. 80% Duodopa + tolcapone

SUMMARY:
The purpose of this study is to determine whether oral intake of COMT inhibitors affects the smooth plasma levodopa levels achieved by intestinal levodopa/carbidopa infusion in advanced Parkinson's disease patients. The hypothesis is that COMT inhibitors make plasma concentrations of levodopa more fluctuating.

DETAILED DESCRIPTION:
The aim is to measure variability in plasma levodopa levels during the following three treatments:

Day 1: Duodopa in individually optimised dose Day 2: 80% of optimised Duodopa dose + two tablets of entacapone at t=0 hours and at t= 6 hours Day 3: 80% of optimised Duodopa dose + two tablets of tolcapone at t=0 hours and at t= 6 hours Plasma samples for determination of levodopa concentrations will be taken every 30 minutes during 8 hours. Video recordings will be performed every 30 min during 8 hours, for later blinded assessments by 2-3 experts. Sequences will be in randomised order. Patient self-scores regarding mobility will be recorded, every 30 min during 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Duodopa treatment ongoing
* Hoehn & Yahr stage 3-5 at worst

Exclusion Criteria:

* Ongoing treatment with COMT inhibitors
* Dementia
* Psychosis
* Treatment with typical neuroleptics
* Contraindications for entacapone or tolcapone

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Difference in coefficient of variation of levodopa in plasma between baseline (day 1) and each of the days on COMT inhibitors. | 3 days

SECONDARY OUTCOMES:
Difference in Treatment Response Scale between the treatments. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Dag Nyholm, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Nyholm D. Enteral levodopa/carbidopa gel infusion for the treatment of motor fluctuations and dyskinesias in advanced Parkinson's disease. Expert Rev Neurother. 2006 Oct;6(10):1403-11. doi: 10.1586/14737175.6.10.1403. PMID 17078781